CLINICAL TRIAL: NCT04739020
Title: Measurement of Respiratory Aerosols in PCR SARS-CoV-2 Positive and Negative Children and Adults
Brief Title: Respiratory Aerosols in Patients With COVID-19 and Healthy Controls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Palas GmbH (Unknown)
Responsible Party: Principal Investigator, Stefan Zielen, Professor Stefan Zielen, Johann Wolfgang Goethe University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-1001
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: SARS-CoV-2 Infection; Covid19
Keywords: COVID-19; Aerosol; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Spirometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PCR SARS-CoV-2 Negative Adults (Active Comparator): Healthy adults with recent negative SARS-CoV-2 PCR test (nasopharyngeal swab). Will consist of parents of participating children and other healthy volunteers.
  Interventions: Diagnostic Test: Resp-Aer-Meter; Diagnostic Test: Spirometry; Diagnostic Test: Qualitative and quantitative virus PCR of respiratory secretions in patients with high aerosol concentrations
- PCR SARS-CoV-2 Positive Adults (Active Comparator): Adults with recent positive SARS-CoV-2 PCR test (nasopharyngeal swab). Will consist of asymptomatic parents that are in the hospital with their children and symptomatic adults that are admitted to the infectious disease ward.
  Interventions: Diagnostic Test: Resp-Aer-Meter; Diagnostic Test: Spirometry; Diagnostic Test: Qualitative and quantitative virus PCR of respiratory secretions in patients with high aerosol concentrations
- PCR SARS-CoV-2 Negative Children (Active Comparator): Children with recent negative SARS-CoV-2 PCR test (nasopharyngeal swab). Will consist of children admitted to the Children's Hospital or presenting for planned diagnostic testing or follow up.
  Interventions: Diagnostic Test: Resp-Aer-Meter; Diagnostic Test: Spirometry; Diagnostic Test: Qualitative and quantitative virus PCR of respiratory secretions in patients with high aerosol concentrations
- PCR SARS-CoV-2 Positive Children (Active Comparator): Children with recent positive SARS-CoV-2 PCR test (nasopharyngeal swab). Will consist of asymptomatic children that are admitted to the Children's Hospital for reasons other than COVID-19 and symptomatic children.
  Interventions: Diagnostic Test: Resp-Aer-Meter; Diagnostic Test: Spirometry; Diagnostic Test: Qualitative and quantitative virus PCR of respiratory secretions in patients with high aerosol concentrations

INTERVENTIONS:
Diagnostic Test: Resp-Aer-Meter — Measurement of respiratory aerosols (particle size and concentration) through breathing into the Resp-Aer-Meter for 3-6 Minutes and comparison between groups.
Diagnostic Test: Spirometry — Comparison of peak expiratory flow (PEF) and forced expiratory volume in one second (FEV1) between groups.
Diagnostic Test: Qualitative and quantitative virus PCR of respiratory secretions in patients with high aerosol concentrations — Comparison between result of aerosol measurement and quantitative and qualitative virus PCR of respiratory secretions that are caught in a filter in which the patient breathes for 10 minutes. Test will be conducted on patients with high aerosol concentrations (>5000/L).

SUMMARY:
The proposed study will investigate respiratory aerosols in SARS-CoV-2 (Severe Acute Respiratory Syndrome Corona Virus 2) positive and negative children and adults with the Resp-Aer-Meter (Palas GmbH). For this purpose, first, the measurement of respiratory aerosols (particle sizes and concentration) with the Resp-Aer-Meter will be established. Thereafter, a comparison between polymerase chain reaction (PCR) SARS-CoV-2 positive and negative participants (children and adults) will be conducted. In addition to the measurement of aerosols, the clinical symptoms, lung function (FEV1) and laboratory inflammatory markers will be analyzed.

DETAILED DESCRIPTION:
Corona virus disease 2019 (COVID-19) is a viral illness caused by SARS-CoV-2. Current research suggests that the SARS-CoV-2 infection is primarily spread through droplets and aerosols. As per current literature, the spread through asymptomatic carriers, as well as highly contagious carriers ('super spreader') play an important role in the infectiousness of the virus. It is currently unclear, if the contagiousness of children differs from adults.

In the proposed investigation, measurement of the particle size and concentration in respiratory aerosols will be conducted via the Resp-Aer-Meter (Palas GmbH). First step will be to establish the measurements with this new device. Thereafter, a comparison between PCR SARS-CoV-2 positive and negative participants, as well as between children and adults, will be conducted. In addition to the measurement of aerosols, the clinical symptoms suggestive of COVID-19, lung function (FEV1) and laboratory inflammatory markers, if available, will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 years or older
* SARS-CoV-2 PCR testing within the last 3 days
* Ability to capture extend and consequences of the study
* Written informed consent of patient and, if applicable, of caregiver

Exclusion Criteria:

* Age under 6 years
* Inability to participate in aerosol measurement
* Inability to participate in Spirometry
* Inability to capture extend and consequences of the study
* Only for arm 1 (PCR SARS-CoV-2 negative adults): chronic disease with immunosuppressive therapy

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Aerosol concentration in PCR SARS-CoV-2 positive and negative participants | Each patient visit will take about 1-2 hours.
  Distinction between PCR SARS-CoV-2 positive and negative participants via aerosol measurement. Especially participants with high aerosol concentrations should be detected.

SECONDARY OUTCOMES:
Change in aerosol concentration over time in PCR SARS-CoV-2 positive participants | 7 days
  Characterization of longitudinal change in aerosol concentration over the course of illness in PCR SARS-CoV-2 positive patients.
Aerosol concentration in children and adults | Each patient visit will take about 1-2 hours.
  Distinction between children and adults via aerosol measurement.
Qualitative and quantitative virus detection in respiratory secretions of patients with high aerosol concentrations. | Each patient visit will take about 1-2 hours.
  Quantitative and qualitative virus PCR measurements of respiratory secretions in participants with aerosol concentrations > 5000/L.
Cofounder Analysis | Each patient visit will take about 1-2 hours.
  Investigation of change in aerosol concentration due to confounders, such as age, sex, other viral illness, lung function, height, weight, BMI and smoking status.
Aerosol concentration and clinical symptoms in PCR SARS-CoV-2 positive participants | Each patient visit will take about 1-2 hours.
  Correlation between clinical symptoms and results of aerosol measurement in PCR SARS-CoV-2 positive participants. Determination if more symptoms lead to higher aerosol concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Professor, Principal Investigator — Johann Wolfgang Goethe University Hospital
Locations (1):
- Johann Wolfgang Goethe University Hospital, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be provided of the investigated cohort
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After end of study, anticipated between June and December 2021
Access Criteria: The data will be available after the end of study and successful publication of the results (anticipated June 2022) for 10 years

REFERENCES:
- [Derived] Gutmann D, Donath H, Herrlich L, Lehmkuhler T, Landeis A, Ume ER, Hutter M, Gossmann AK, Weis F, Weiss M, Rabenau HF, Zielen S. Exhaled Aerosols in SARS-CoV-2 Polymerase Chain Reaction-Positive Children and Age-Matched-Negative Controls. Front Pediatr. 2022 Jul 18;10:941785. doi: 10.3389/fped.2022.941785. eCollection 2022. PMID 35923787